CLINICAL TRIAL: NCT02306564
Title: Effect of Cabergoline on Subendometrial Vascularity During ICSI Cycles and Pregnancy Outcome
Brief Title: Effect of Cabergoline on Endometrial Vascularity During IntraCytoplasmic Sperm Injection
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed M.Kamel, Lecturer of Obstetric & Gynecology, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: A14022014
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Infertility
Keywords: ICSI; cabergoline; Subendometrial vascularity
MeSH Terms: conditions — Infertility | interventions — Cabergoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (Experimental): Group A will include patients at risk of OHSS receiving Cabergoline 0.5mg daily for 8 days (Dostinex®, Pfizer Australia Pty Ltd ) from the day of oocyte pick up for prevention of hyperstimulation
  Interventions: Drug: Cabergoline
- Group B (No Intervention): Group B will include patients AT RISK of ovarian hyperstimulation syndrome (OHSS) not receiving Cabergoline.
- Group C (No Intervention): Group C will serve as a control group and will include age & BMI matched patients NOT AT RISK of OHSS, and not receiving cabergoline.

INTERVENTIONS:
Drug: Cabergoline — given to patients at high risk for OHSS
  Other Names: dostinex
  Arms: Group A

SUMMARY:
The purpose of this study is to determine the effect of giving cabergoline to patients at risk of OHSS (ovarian hyperstimulation syndrome) after ovum pick up, on endometrial vascularity and it's effect on pregnancy outcome

DETAILED DESCRIPTION:
Following ethical approval of the committee of obstetrics & gynecology IVF department of kasr al-Aini hospital Cairo University, 150 women attending the IVF unit of Kasr el Aini hospital for management of infertility will be included in the study after obtaining informed consent from each patient. All women are scheduled for intracytoplasmatic sperm injection (ICSI) after controlled ovarian stimulation.

All women included in the study, after applying eligibility criteria , will be subjected to careful history taking and general and local examination, follicle stimulating hormone (FSH), luteinizing hormone (LH), Antral follicle count (AFC) &Antimullerian hormone (AMH) will be recorded and body mass index (BMI) calculation is done.

BMI is defined as weight in kilograms divided by height in meters squared (kg/m2), Excess weight is BMI ≥ 25 kg/m2 and obesity is BMI ≥ 30 kg/m2.

As most patients needing cabergoline for prevention of hyperstimulation are obese, therefore only those with BMI ≥ 30 kg/m2 will be included in the study. The study will include three groups, each group containing 50 patients.

Group A will include patients at risk of OHSS receiving Cabergoline 0.5mg daily for 8 days (Dostinex®, Pfizer Australia Pty Ltd ) from the day of oocyte pick up for prevention of hyperstimulation. Group B will include patients at risk of ovarian hyperstimulation syndrome (OHSS) not receiving Cabergoline. While group C will serve as a control group and will include age & BMI matched patients not at risk of OHSS, and not receiving cabergoline.

Risk of developing ovarian hyperstimulation syndrome (OHSS) and expectation of high oocyte yield will include serum E2>3,500 pg/ml and more than 20 follicles ≥11 mm on the day of final oocyte maturation, & Patients who underwent coasting for OHSS prevention.

The standard long gonadotrophin-releasing hormone (GnRH) agonist protocol will be used for patients with predicted normal response based on clinical & hormonal profile ; 1 mg of leuprolide acetate daily subcutaneous injection (s.c) (Lucrin ®; Abbott, Hoofddorp, The Netherlands) is applied from the mid luteal phase onward till the day of HCG injection.

Gonadotropins in the form of human menopausal gonadotropin (HMG) (Merional ®, IBSA, Institute Biochimique SA, Lugano, Switzerland) will be given by intramuscular injection (IM) from the 2nd day of menstruation after confirmed down regulation (E2<50pg/ml), The starting dose range from 150 to 300 IU depending on the basal FSH level, AFC, maternal age and BMI.

Patients with high predicted high response as evidenced by high serum AMH (more 4.0 ng/ml), or inverted FSH:LH ratio (polycystic ovarian syndrome PCOS) or, high antral follicle count (over 30) will be given Antagonist protocol where human menopausal gonadotropin (HMG) (Merional ®, IBSA, Institute Biochimique SA, Lugano, Switzerland) will be given IM from the 2nd day of menstruation, The starting dose range from 150 to 300 IU and Gnrh Antagonist cetrorelix acetate (Cetrotide®, Zentaris IVF GmbH, Australia), 0.25 mg S.C, onwards will be given daily when the lead follicle reaches 14mm.

In all protocols, stimulation is monitored by trans-vaginal ultrasonography and serial E2 measurements starting from day 7 of the cycle and the gonadotropin dose is adjusted individually according to follicular response.

After the development of at least three leading follicles≥18 mm, 10,000 unit of HCG (Choriomon, IBSA, Institute Biochimique SA) is given IM, and a trans vaginal ultrasound-guided oocyte retrieval is performed 36 hours later.

Patients with expected high oocyte yield, will be sent on the last day of folliculometry to do three dimensional (3D) power Doppler to determine endometrial vascularity.

After ovum pick up, Oocytes are then fertilized in vitro using ICSI and after three to five days embryo transfer will be done using labotec catheter (Labotec, Gottingen Germany) with ultrasound guidance.

A second Trans-vaginal U/S demonstrating endometrial vascularity will be done 1 hour before embryo-transfer.

Progesterone pessaries 400 mg twice daily (Cyclogest 400mg ®Actavis plc. Dublin, Ireland) is given as a luteal support starting from the day of embryo transfer and continued for 16 days after.

Pregnancy is defined as the occurrence of a positive beta human chorionic gonadotrophin (βHCG) >10 IU on day 12 after embryo transfer and a second higher value 2 days later, followed by ultrasonography confirmation of cardiac activity at 6 weeks gestation.

The criteria for cycle cancellation are:

* The presence of less than three follicles.
* E2 level less than500 pg/ml.

All 3D ultrasound and power Doppler examinations will be carried out by one investigator on the day of final oocyte maturation and repeated again on the day of embryo transfer, 1 hour before the procedure.

The Voluson 730 machine (GE Healthcare Austria GmbH, Seoul, Korea) with an endocavitary volumetric 4-9MHz vaginal probe after bladder evacuation, Computer-Aided Analysis (VOCAL™) Imaging Program for the 3D power Doppler histogram analysis will be used to measure the endometrial volume (EV) and 3D power Doppler indices within the endometrium .

Vascularization index (VI) measures the ratio of the number of color voxels to the total number of voxels (%) and represents the presence of blood vessels (vascularity). Flow index (FI) measures the mean power Doppler signal intensity (0-100) and represents the average intensity of blood flow. Vascularization flow index (VFI) is calculated by multiplying VI and FI (0-100) and represents a combination of vascularity and flow intensity

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 - ≤40 years
2. Normal serum prolactin level.
3. Tubal factor of infertility.
4. Unexplained infertility.
5. BMI ≥ 30 kg/m2.
6. Estradiol (E2)>3,500 pg/ml on day of ovulation trigger.
7. Patients who underwent coasting for OHSS prevention.
8. More than 20 follicles ≥11 mm on the day of final oocyte maturation.

Exclusion criteria:

1. Contraindication of pregnancy e.g.: Somatic and mental diseases, which are contraindications for carrying of a pregnancy and childbirth, inborn malformations or acquired deformations of uterus cavity which make embryo implantation or carrying of a pregnancy impossible ,ovarian tumors.
2. Severe Male factor infertility.
3. Hyperprolactinemic patients.
4. Frozen embryo transfer cycles
5. Uterine Anomalies.
6. Uterine synechia.
7. History of Genital Tuberculosis.
8. Repeated implantation failure in ICSI.
9. On medication that is known to alter prolactin levels e.g antipsychotics, Atypical agents and risperidone
10. Thyroid dysfunction.
11. Medical disorders affecting serum prolactin eg acromegaly ,chronic renal failure and hypothyroidism

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-11 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate (chemical , clinical). | 2 weeks after embryo transfer
  beta human chorionic gonadotrophin (βHCG) >10 IU on day 12 after embryo transfer

SECONDARY OUTCOMES:
Miscarriage rate | 3 weeks after positive βHCG
  first ultrasound at 7 weeks gestation
OHSS rate | 4 weeks
  early and late onset OHSS
Vascularization index (VI) | 5 days
  3D ultrasound and power Doppler examination done before ovum pick up and repeated before transfer
Flow index (FI) | 5 days
  3D ultrasound and power Doppler examination done before ovum pick up and repeated before transfer
vascularization flow index (VFI) | 5 days
  3D ultrasound and power Doppler examination done before ovum pick up and repeated before transfer
pulsatility index (PI) | 5 days
  3D ultrasound and power Doppler examination done before ovum pick up and repeated before transfer
the resistance index (RI) | 5 days
  3D ultrasound and power Doppler examination done before ovum pick up and repeated before transfer
the peak systolic velocity (Vp). | 5 days
  3D ultrasound and power Doppler examination done before ovum pick up and repeated before transfer
the end-diastolic velocity (Vd). | 5 days
  3D ultrasound and power Doppler examination done before ovum pick up and repeated before transfer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Kamel, MD, Principal Investigator — Lecturer of obstetrics & Gynecology
Locations (1):
- Assissted reproduction unit Kasr alaini hospital, Ḩadā’iq al Qubbah, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Tang H, Mourad SM, Wang A, Zhai SD, Hart RJ. Dopamine agonists for preventing ovarian hyperstimulation syndrome. Cochrane Database Syst Rev. 2021 Apr 14;4(4):CD008605. doi: 10.1002/14651858.CD008605.pub4. PMID 33851429